CLINICAL TRIAL: NCT06954142
Title: Restricted Versus Liberal Fluid Intake for Prevention of Bronchopulmonary Dysplasia - RELIEF Trial. A Cluster-randomised Multiple Period Cross-over Trial.
Brief Title: Restricted Versus Liberal Fluid Intake for Prevention of Bronchopulmonary Dysplasia
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss Neonatal Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-00321; ks22Schulzke
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Fluid Restriction; Preterm Infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Pragmatic, registry-linked, multicentre, open-label, cluster-randomised, multiple period, cross-over, effectiveness trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction (Experimental): Fluid restriction strategy (fluid target 135 ±5 mL/kg/d). This is standard of care.
  Interventions: Other: Fluid restriction
- Liberal fluid intake (Active Comparator): Liberal fluid intake strategy (fluid target 165 ± 5 mL/kg/d) in line with international best practice recommendations on nutrition.
  Interventions: Other: Liberal fluid intake

INTERVENTIONS:
Other: Fluid restriction — Fluid restriction strategy (fluid target 135 ±5 mL/kg/d)
  Arms: Fluid restriction
Other: Liberal fluid intake — Liberal fluid intake strategy (fluid target 165 ± 5 mL/kg/d)
  Arms: Liberal fluid intake

SUMMARY:
The aim of this study is to determine whether restricted fluid intake (135 ±5 mL/kg/day) compared to liberal fluid intake (165 ±5 mL/kg/day) from day 8 of life reduces the incidence of bronchopulmonary dysplasia (BPD) at 36 weeks postmenstrual age or prior death in preterm infants born <30 weeks gestational age.

DETAILED DESCRIPTION:
Complications of preterm birth remain the leading cause of death in children under five years of age worldwide, accounting for approximately one million deaths annually. Among the survivors, bronchopulmonary dysplasia (BPD) is the most common severe complication. BPD is a chronic lung disease characterized by prolonged need for respiratory support and oxygen therapy, poor postnatal growth, and long-term impairments in lung function and neurodevelopment.

Despite advancements in neonatal care, BPD is the most common chronic lung disease in infancy and associated with increased mortality, repeated hospitalisation throughout childhood, impaired lung function up into adulthood, and long-term neurodevelopmental impairment. The incidence of BPD has remained stable over the past 15 years. This is likely due to the improved survival of extremely preterm infants, who are at the highest risk for BPD.

A key feature of evolving BPD is the accumulation of interstitial pulmonary edema, which reduces lung compliance and increases the need for respiratory support, thereby perpetuating a cycle of lung damage.

Currently, diuretics are sometimes used to manage pulmonary edema in preterm infants. While they can improve lung function in the short term, they come with potential risks including bone demineralization, nephrotoxicity, electrolyte imbalances, and impaired growth.

As a potentially safer alternative, fluid restriction is sometimes used to prevent or manage pulmonary edema. It is hypothesized to improve lung mechanics and reduce the need for respiratory support, without the adverse effects associated with medications. However, there is no robust evidence on optimal fluid targets in these patients.

SwissNeoNet, consisting of all nine Swiss NICUs, is a mandatory national registry, where data on all infants born before 32 weeks of gestation and/or with a birth weight < 1501 g are collected. Fluid management practices vary among Swiss neonatal intensive care units (NICUs) following international guidelines recommending 135 to 180 mL/kg/day of fluids. This variation may contribute to the differing rates of BPD and mortality observed across centers, but fluid intake is not routinely captured in SwissNeoNet data, making it difficult to assess its impact.

In summary, although fluid restriction shows potential as a simple and low-risk intervention to reduce the incidence of BPD, current evidence is insufficient to support its routine use. There is a clear need for a robust, contemporary, and pragmatic trial to evaluate whether fluid restriction, started after the first week of life, can safely and effectively reduce the incidence of BPD or death in very preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised preterm infants born before 30 weeks 0 days gestation
* Signed informed consent for further research use of health-related data

Exclusion Criteria:

* congenital malformations
* diseases likely to affect life expectancy, lung function, fluid strategy, or neurodevelopment
* renal disease requiring fluid management outside the clinical standard of care
* congenital heart disease not including patent ductus arteriosus (PDA)

Min Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia (BPD) | From enrolment to 36 weeks postmenstrual age
  Proportion of infants with BPD measured at 36 weeks postmenstrual age or prior death.

SECONDARY OUTCOMES:
Complications of prematurity | From enrolment to 36 weeks postmenstrual age
  Major complications of prematurity including necrotising enterocolitis ≥ Bell's stage 2, retinopathy of prematurity requiring treatment, patent ductus arteriosus requiring treatment, abnormal brain ultrasound, late onset sepsis
Days to reach full feeds | From enrolment to 36 weeks postmenstrual age
  Days to reach full feeds defined as 150 ml/kg/d or being off parenteral nutrition
Need of diuretics | From enrolment to 36 weeks postmenstrual age
  Treatment with diuretics (days on diuretics)
Need of corticosteroids | From enrolment to 36 weeks postmenstrual age
  Systemic postnatal corticosteroids for prevention or treatment of bronchopulmonary dysplasia
Need of respiratory support | At first discharge home, on average 37 weeks postmenstrual age
  Duration of mechanical ventilation, non-invasive respiratory support, total positive pressure support, supplemental oxygen support, supplemental home oxygen, home ventilation
Growth | at birth and 36 weeks postmenstrual age
  difference in weight, length, and head circumference z-score at 36 weeks postmenstrual age and at birth, respectively
Daily caloric intake | From enrolment to 36 weeks postmenstrual age
  Daily caloric intake from day 8 of life to 36 weeks postmenstrual age
Dehydration | From enrolment to 36 weeks postmenstrual age
  Dehydration (sodium level ≥ 150 mmol/L plus clinical signs of dehydration)
Fluid overload | From enrolment to 36 weeks postmenstrual age
  Fluid overload (sodium level ≤ 130 mmol/L plus clinical signs of fluid overload)
Age at discharge | At first discharge home, on average 37 weeks postmenstrual age
  Postmenstrual age at discharge home
Tube feeding | At first discharge home, on average 37 weeks postmenstrual age
  Tube feeding at discharge home

OTHER OUTCOMES:
Growth | from 36 weeks postmenstrual age, 6-12 and 18-24 months post-term
  Growth (weight, length, and head circumference z-score)
Respiratory outcome | from 36 weeks postmenstrual age, 6-12 and 18-24 months post-term
  Respiratory outcome as per Basel-Bern-Infant-Lung-Development cohort study questionnaire
Visits to the emergency | From discharge to 6-12 and 18-24 months
  Visits to the emergency department from discharge to 6-12 months for any reason
Neurodevelopmental outcome | from enrolment to 18-24 months post-term
  Neurodevelopmental outcome as per PARCA-R questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schulzke, Prof.MD, Principal Investigator — University Children's Hospital Basel, UKBB
Locations (9):
- Switzerland (9):
  - Kantonsspital Aarau AG, Klinik für Kinder u. Jugendliche, Aarau
  - University Children's Hospital Basel (UKBB), Basel
  - Inselspital Bern, Kinderklinik, Bern
  - Kantonsspital Graubünden, Departement Kinder- und Jugendmedizin, Chur
  - Hôpitaux universitaires de Genève (HUG), Unité de Néonatologie, Geneva
  - Centre hospitalier universitaire vaudois (CHUV) - Service de néonatologie, Lausanne
  - Luzerner Kantonsspital, Kinderspital, Lucerne
  - Ostschweizer Kinderspital & Neonatologie und Frauenklinik KSSG, Perinatalzentrum St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Klinik für Neonatologie, Zurich